CLINICAL TRIAL: NCT04299451
Title: The Efficacy of Open Dialogue About Complementary Alternative Medicine Integrated in Conventional Oncology Care. Patient Reported Quality of Life and Well-being (CAMONCO 2)
Brief Title: Open Dialogue About Complementary Alternative Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAMONCO 2
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Cancer
Keywords: Alternative Medicine; Cancer; Communication; Complementary medicine; Dialogue; Integrative medicine; Oncology
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open dialogue about CAM (ODC-COC) (Experimental): Participation in an open dialogue about CAM with a nurse specialist. The dialogue will be based on the fundamentals of person-centered care and include patient preferences and wishes, reliable information and counselling, and advice about the potential risks and benefits of using CAM.
  The dialogue is estimated to last approximately 60 minutes and all dialogues will be conducted by the same nurse. Depending on patient needs and wishes there may be a follow-up consultation one month after the first dialogue.
  Interventions: Other: Open dialogue about CAM
- Standard care (No Intervention): Standard care including referral to a homepage about complementary alternative medicine

INTERVENTIONS:
Other: Open dialogue about CAM — 1-hour dialogue about CAM with a nurse specialist as an integrated part of conventional oncology care
  Arms: Open dialogue about CAM (ODC-COC)

SUMMARY:
The purpose of this phase III parallel-group randomized controlled trial is to assess the efficacy of open dialogue about complementary alternative medicine integrated in conventional oncology care (ODC-COC). The investigators hypothesize that patients in the intervention group participating in an ODC-COC with a nurse specialist report better quality of life compared to patients in the control group receiving standard care alone.

DETAILED DESCRIPTION:
Patients randomized to the intervention group will participate in a scheduled ODC-COC with a specialist nurse, who has completed the Fellowship in Integrative Medicine at the University of Arizona. This is a training program for health professionals in empowering individuals and communities to optimize health and well-being through evidence-based, sustainable and integrative approaches. The ODC-COC will be based on the fundamentals of person-centered care according to this program and include patient preferences and wishes, reliable information and counselling and advice about the potential risks and benefits of using complementary alternative medicine as an adjunct to conventional oncology care.

The dialogue lasts approximately 60 minutes and will take place as soon as possible and no later than two weeks after enrolment. The same nurse will conduct all dialogues. According to patient needs and wishes there may be a follow-up dialogue over the telephone or in the Oncology Outpatient Clinic. The potential second dialogue is estimated to last approximately 30 minutes.

Participants in the control group will receive standard information including reference to www.KABcancer.dk, which is a website presenting research on CAM, including information about its potential effects and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and reads Danish
* Diagnosed with a new primary cancer or a relapse of cancer within the last 3 months
* Planned or initiated medical oncology treatment at the Department of Oncology, Vejle Hospital
* At least two months of oncology treatment is realistic based on clinical assessment
* Life expectancy of at least six months
* Informed consent

Exclusion Criteria:

-Participation in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in patient reported quality of life between the two arms at 8 weeks as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ CAT core) | 8 weeks after enrollment
  This instrument lists individually tailored questions assessing quality of life, including functional scales, symptom scales, global health status, and psychosocial scales.

SECONDARY OUTCOMES:
Difference in patient reported quality of life between the two arms at 12 and 24 weeks as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ CAT Core). | At baseline and after 12 and 24 weeks
  This instrument lists individually tailored questions assessing quality of life, including functional scales, symptom scales, global health status, and psychosocial scales.
Difference in patient reported level of depression and anxiety between the two arms as measured by the Hospital Anxiety and Depression Scale (HADS). | At baseline and 8, 12 and 24 weeks after enrollment
  With 14 questions this instrument assesses the symptom severity and caseness of anxiety disorders and depression.
Difference in patient reported top concerns in the two arms as measured by the Measure Yourself Concerns and Wellbeing (MYCaW) questionnaire. | At baseline and 8, 12 and 24 weeks after enrollment
  This instrument assesses the level of severity of the two most pressing concerns and present overall well-being
Difference in patient reported decision regret in the two arms as measured by the Decision Regret Scale (DRS). | At baseline and 8 weeks after enrollment
  This instrument consists of 5 items elucidating if regret is present, whether the decision is the right one, and whether the patient would make the same decision again.
Difference in overall survival between the two arms | 12 months after enrollment of last patient
  Kaplan-Meier survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henrik Jensen, MD, PhD, Study Chair — Department of Oncology, Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stie M, Delmar C, Norgaard B, Jensen LH. Efficacy of open dialogue about complementary and alternative medicine compared with standard care in improving quality of life in patients undergoing conventional oncology treatment (CAMONCO 2): protocol for a randomised controlled trial. BMJ Open. 2022 Apr 25;12(4):e059960. doi: 10.1136/bmjopen-2021-059960. PMID 35470199